CLINICAL TRIAL: NCT06924554
Title: Study Protocol of a Non-randomized Controlled Trial on a Circumplex Model-based Motivational Training Program for Pre-service Physical Education Teachers
Brief Title: Motivational Training Program for Pre-service Physical Education Teachers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Carlos Mayo Rota, Principal Investigator, Universidad de Zaragoza
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PROYS01_24
Record Dates: First submitted 2025-03-21; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Teaching Styles; Motivation; Competence; Pre-service Teachers
Keywords: Self-Determination Theory; (de)motivating teaching styles; physical education teacher education; quasi-experimental study; mixed-methods research

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group will participate in a 14-hour training program combining theoretical and practical components of Self-Determination Theory and the circumplex model.
  Interventions: Behavioral: Motivational Training Program
- Control group (No Intervention): The control group will follow the standard Physical Education Teacher Education curriculum

INTERVENTIONS:
Behavioral: Motivational Training Program — This study presents the protocol for a non-randomized controlled trial evaluating a motivational-based training program for pre-service Physical Education teachers, grounded in Self-Determination Theory and the circumplex model. The program, embedded in a Master's in Physical Education Teacher Education, consists of theoretical and practical training to foster motivating teaching styles and minimize demotivating ones. The study will involve at least 38 pre-service teachers, divided into an experimental group (n = 19) and a control group (n = 19). The experimental group will participate in a 14-hour training program combining theoretical and practical components. The control group will follow the standard Physical Education Teacher Education curriculum.
  Arms: Experimental group

SUMMARY:
This study presents the protocol for a non-randomized controlled trial evaluating a motivational-based training program for pre-service Physical Education teachers. The experimental group will participate in a 14-hour training program based on Self-Determination Theory and the circumplex model. The program consists of theoretical and practical training to foster motivating teaching styles and minimize demotivating ones. The control group will follow the standard curriculum of the Master's in Physical Education Teacher Education program without exposure to the specific intervention.

DETAILED DESCRIPTION:
Physical Education Teacher Education is crucial, as it directly influences how pre-service Physical Education teachers will teach, motivate, and engage their future students. However, training programs that foster motivating teaching styles while minimizing demotivating ones remain scarce, particularly during initial teacher education. This study presents the protocol for a non-randomized controlled trial evaluating a motivational-based training program for pre-service Physical Education teachers, grounded in Self-Determination Theory and the circumplex model. The program, embedded in a Master's in Physical Education Teacher Education, consists of theoretical and practical training to foster motivating teaching styles and minimize demotivating ones. The study will involve at least 38 pre-service teachers, divided into an experimental group (n = 19) and a control group (n = 19). The experimental group will participate in a 14-hour training program combining theoretical and practical components. The control group will follow the standard Physical Education Teacher Education curriculum. A quasi-experimental pre-post design with a mixed-methods approach will be used. Quantitative assessments will measure changes in perceived competence, motivation for teaching, and (de)motivating teaching styles, while qualitative focus groups will provide in-depth insights into participants' experiences and program applicability. To ensure objectivity, independent researchers will conduct assessments, and external experts will moderate the focus groups. Findings will contribute empirical evidence on the effectiveness of Self-Determination Theory-based interventions in initial teacher education, informing curriculum development and supporting the advancement of evidence-based pedagogical training in Physical Education.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in the Master's in Physical Education Teacher Education at the University of Zaragoza.
* 100% attendance in training sessions (experimental group).
* Completion of questionnaires at three time points (pre-test, intermediate, and post-test).
* Participation in the final focus group discussion.

Exclusion Criteria:

* Failure to complete required assessments.
* Lack of attendance in mandatory sessions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
(De)motivating teaching styles | At baseline (Week 0), 4 weeks after baseline, and 8 months after baseline.
  Changes in (de)motivating teaching styles (Measured using SIS-PE)
Teaching competence | At baseline (Week 0), 4 weeks after baseline, and 8 months after baseline.
  Changes in perceived teaching competence (Measured using BPNSFS).
Motivation to teach | At baseline (Week 0), 4 weeks after baseline, and 8 months after baseline.
  Changes in motivation to teach (Measured using EME-ES).

SECONDARY OUTCOMES:
Quality of the training program | 4 weeks after baseline, and 8 months after baseline.
  Perceived quality of the training program (Program evaluation questionnaire and final focus group).
Applicability of the training program | 4 weeks after baseline, and 8 months after baseline.
  Perceived applicability of the training program (Program evaluation questionnaire and final focus group).
Strengths and weaknesses of the training program | 8 months after baseline.
  Qualitative insights on the impact of the training (Final focus group discussion)

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad de Ciencias Humanas y de la Educación, Huesca, Aragon, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mayo-Rota C, Abos A, Garcia-Cazorla J, Villafana-Samper Z, Garcia-Gonzalez L. Study protocol of a non-randomized controlled trial on a circumplex model-based motivational training program for pre-service physical education teachers. Front Public Health. 2025 Jul 7;13:1611556. doi: 10.3389/fpubh.2025.1611556. eCollection 2025. PMID 40692882

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-20): https://cdn.clinicaltrials.gov/large-docs/54/NCT06924554/Prot_SAP_000.pdf